CLINICAL TRIAL: NCT06284057
Title: Double Kissing (DK) vs Culotte Culotte. Lower Silesia Culotte Bifurcation Registry (LSCBR).
Brief Title: Lower Silesia Culotte Bifurcation Registry (LSCBR).
Acronym: LSCBR
Status: Recruiting | Type: Observational
Sponsor: Regional Cardiology Center, The Copper Health Centre (MCZ), (Other)
Collaborators: Department of Cardiology, Provincial Specialized Hospital in Legnica, 59-200 Legnica, Poland. (Unknown)
Responsible Party: Principal Investigator, Adrian Włodarczak, Professor, Regional Cardiology Center, The Copper Health Centre (MCZ),
Other Study IDs: CopperHealthCentre3
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Safety Issues; Efficacy, Self
Keywords: Percutaneous coronary intervention (PCI); Bifurcation lesion; Culotte Technique; Double Kiss Culotte Technique; Acute Coronary Syndrome; Two-Stent Technique
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Culotte Group: Data regarding patient with performed PCI- bifurcation with subsequent implantation of two stents using the Culotte technique
  Interventions: Procedure: Bifurcation PCI with two stent technique Culotte Technique or Double Kiss (DK) Culotte
- Double Kiss (DK) Culotte Group: Data regarding patient with performed PCI- bifurcation with subsequent implantation of two stents using the Double Kiss- Culotte technique. DK-Culotte technique is a variety of classical "Culotte techniques" in which one additional kissing balloon dilation is performed just after SB stenting, and prior to MB stent implantation.
  Interventions: Procedure: Bifurcation PCI with two stent technique Culotte Technique or Double Kiss (DK) Culotte

INTERVENTIONS:
Procedure: Bifurcation PCI with two stent technique Culotte Technique or Double Kiss (DK) Culotte — Patient with CAD and coexisting bifurcation lesion requiring two-stent approach treated with Culotte Technique or Double Kiss (DK) Culotte due to operator distraction.

SUMMARY:
The study aimed to evaluate the outcomes of bifurcation PCI using two techniques (Culotte vs. DK-Culotte) using data from a retrospective analysis.

DETAILED DESCRIPTION:
The study contains a retrospective analysis of subjects who have undergone PCI in two high-volume cooperative Cardiac Departments in the Lower Silesia Region (Poland) between April 2012 and January 2024. Data regarding all performed PCI from these periods were prescreened in terms of bifurcation lesion with subsequent implantation of two stents using the Culotte technique or the DK-Culotte technique. The indication for percutaneous coronary intervention (PCI) was based either on a judgment made by the Heart Team or on a particular clinical indication (ongoing ischemia, lack of will for the alternative treatment options, presence of significant angiographic CAD suitable for PCI due to ESC/ESH recommendation). The decision to perform the two-stent technique PCI was left to the operator's dissertation based on clinical and angiographical features. All patients were thoroughly informed about all therapeutic options and PCI-related risks before providing written informed consent for the procedure. There were no clinical or vessel-related exclusion criteria (lesion anatomy, length, tortuosity, severity). However, patients who had undergone PCI with coronary stents prior to the index procedure with respect to the bifurcation lesion studied were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Presence of significant changes in the coronary bifurcation requiring the implantation of two coronary stents using the Culotte or DK Culotte technique.

Exclusion Criteria:

* Patients who underwent PCI with coronary stents prior to the index procedure for the bifurcation lesion studied.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study includes a retrospective analysis of subjects who underwent PCI in two cooperative cardiac centers in the Lower Silesia region between April 2012 and January 2024. Data from the participating centers on all PCIs performed during these periods were prescreened for bifurcation lesions with subsequent implantation of two stents using the Culotte technique or the DK-Culotte technique. The indication for percutaneous coronary intervention (PCI) was based on the judgment of the cardiac team or on a specific clinical indication (persistent ischemia, unwillingness to accept alternative treatment options, presence of significant angiographic CAD suitable for PCI). The decision to perform PCI with the two-stent technique was left to the operator's judgment based on clinical and angiographic characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-04-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Target lesion failure (TLF) | Final assessment - 5 years after the initial hospitalization; followed by evaluation every 6 months from the end of the hospitalization until the final assessment (5 years)
  The primary endpoint was target lesion failure (TLF): the composite of cardiac death, target vessel myocardial infarction (TVMI), or clinically driven TLR.

SECONDARY OUTCOMES:
MACE | Final assessment - 5 years after the initial hospitalization; followed by evaluation every 6 months from the end of the hospitalization until the final assessment (5 years)
  The secondary composed outcome was MACE: myocardial infarction (MI), cardiac death, MB-TLR or/and SB-TLR

OTHER OUTCOMES:
Stent thrombosis | Final assessment - 5 years after the initial hospitalization; followed by evaluation every 6 months from the end of the hospitalization until the final assessment (5 years)
  Stent thrombosis in a stent implanted in a bifurcation during primary intervention. Stent thrombosis was defined according to The Academic Research Consortium-2 consensus document.
  The presence of a thrombus† that originates in the stent/scaffold or in the segment 5 mm proximal or distal to the stent/scaffold or in a side branch originating from the stented/scaffolded segment and the presence of at least 1 of the following criteria:
  1)Acute onset of ischemic symptoms at rest 2)New electrocardiographic changes suggestive of acute ischemia 3)Typical rise and fall in cardiac biomarkers (refer to definition of spontaneous myocardial infarction) or Pathological confirmation of stent/scaffold thrombosis
Stent restenosis | Final assessment - 5 years after the initial hospitalization; followed by evaluation every 6 months from the end of the hospitalization until the final assessment (5 years)
  Stent restenosis in a stent placed in a bifurcation during primary intervention. Stent restenosis should be confirmed by either angiography or intravascular assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Włodarczak, Assoc. Prof., Principal Investigator — Regional Cardiology Center, The Copper Health Centre (MCZ),
Locations (2):
- Poland (2):
  - Department of Cardiology, Provincial Specialized Hospital in Legnica,, Legnica, Lower Silesian Voivodeship
  - Department of Cardiology, The Copper Health Centre (MCZ), Lubin, Lower Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: Undecided